CLINICAL TRIAL: NCT00080262
Title: Phase II Study of Novel Epothilone (BMS-247550) in Patients With MBC Who Are Refractory to an Anthracycline, a Taxane, and Capecitabine
Brief Title: Novel Epothilone (BMS-247550) in Patients With Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-081
Record Dates: First submitted 2004-03-25; First posted 2004-03-26 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Metastases
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — ixabepilone

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Solution, IV, 40 mg/m2, every 21 days, extended, until PD or discontinued for other reasons.
  Other Names: BMS-247550

SUMMARY:
The purpose of this research study is to assess the response rate of the investigational drug BMS-247550 (Ixabepilone) in women with metastatic breast cancer who are refractory to an anthracycline, a taxane, and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received all 3 drugs- an anthracycline, taxane, and capecitabine (alone or in combination) and be resistant
* No more than 3 prior chemotherapy regimens in the metastatic setting
* Must have at least one target lesion that is radiographically measurable
* Good performance status
* No history of or current brain or leptomeningeal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Response rate as determined by the IRRC

SECONDARY OUTCOMES:
Time to progression, duration of response, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (17):
  - Local Institution, La Verne, California
  - Local Institution, Meriden, Connecticut
  - Local Institution, Jacksonville, Florida
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, New York, New York
  - Local Institution, Asheville, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Jackson, Tennessee
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
- Argentina (2):
  - Local Institution, Buenos Aires
  - Local Institution, Santa Fe
- Local Institution, Montreal, Quebec, Canada
- France (7):
  - Local Institution, Besançon
  - Local Institution, Bobigny
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (2):
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt Hoechst
- Mexico (3):
  - Local Institution, Mérida, Yucatán
  - Local Institution, Chihuahua City
  - Local Institution, Distrito Federal
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Trondheim
- South Africa (5):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Fichardtpark, Free State
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Overport, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- Sweden (4):
  - Local Institution, Helsingborg
  - Local Institution, Lund
  - Local Institution, Malmo
  - Local Institution, Stockholm

REFERENCES:
- [Background] Perez EA, Lerzo G, Pivot X, Thomas E, Vahdat L, Bosserman L, Viens P, Cai C, Mullaney B, Peck R, Hortobagyi GN. Efficacy and safety of ixabepilone (BMS-247550) in a phase II study of patients with advanced breast cancer resistant to an anthracycline, a taxane, and capecitabine. J Clin Oncol. 2007 Aug 10;25(23):3407-14. doi: 10.1200/JCO.2006.09.3849. Epub 2007 Jul 2. PMID 17606974